CLINICAL TRIAL: NCT03259828
Title: Interfraction and Intrafraction Organ Motion of the Sigmoid Colon in Patients With Colorectal Cancer Undergoing Adjuvant Radiotherapy
Brief Title: Sigmoid Colon Organ Motion in Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Tsai, Mu-Hung, Attending Physician, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-106-037
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Sigmoid Cancer; Sigmoid Colon Cancer
Keywords: Sigmoid colon cancer; Internal organ motion; Radiotherapy
MeSH Terms: conditions — Sigmoid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant image-guided radiotherapy (Experimental): Adjuvant radiotherapy with image guidance via cone beam computed tomography. Treatment is identical to the current standard of care.
  Interventions: Radiation: Adjuvant image-guided radiotherapy

INTERVENTIONS:
Radiation: Adjuvant image-guided radiotherapy — Image-guided adjuvant radiotherapy to the sigmoid colon surgical tumor bed and pelvic regional lymph nodes: 45-50.4 Gy in 1.8 Gy/fraction

SUMMARY:
Radiotherapy is used in cancer treatment to eradicate microscopic cancer cells to lower the risk of recurrence. The radiotherapy plan must account for organ movement inside the body to ascertain adequate dose is delivered to the target. Knowledge of the magnitude is crucial to radiotherapy treatment planning. This study aims to quantify the movement of the sigmoid colon between different fractions of radiotherapy treatment (interfraction motion) and within the same fraction (intrafraction motion). This knowledge will help us determine the optimal margin to use in radiotherapy treatment planning.

DETAILED DESCRIPTION:
Day-to-day positioning variations contribute to uncertainty in radiotherapy. The International Commission on Radiation Units and Measurements (ICRU) report 62 recommended a margin added to the clinical target volume (CTV) to produce the planning target volume (PTV). In ICRU report 83, this concept is further extended and refined to yield the internal target volume (ITV), which is defined as CTV plus a margin to account for uncertainty within the patient. Image-guided radiotherapy (IGRT) has been developed as a method to lower the margin required in PTV expansion. In current practice, IGRT methods mostly rely on bony anatomy alignment. Due to its nature, internal organ motion cannot be compensated by IGRT. Therefore, an ITV expansion is still required. The optimal ITV expansion margin depends on the magnitude of internal organ motion; the smallest margin that provides adequate coverage is preferred.

In this study, we aim to quantify organ motion of the sigmoid colon anastomosis site during radiotherapy treatment, including movement between fractions (interfraction) and movement within the same fraction (intrafraction).

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed sigmoid colon cancer, who have received surgical excision (AR or LAR).
* Anastomosis of the colon must be performed with a surgical stapler, with the staple visible on CT imaging.

Exclusion Criteria:

* Gross recurrent disease (defined as visible mass on CT imaging) in the pelvis.
* Other malignancy within the pelvic cavity.
* Previous surgery to the pelvic cavity other than AR/LAR.
* Pregnant or lactating females.
* Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Interfraction sigmoid colon organ motion | 90 days
  Offset of the sigmoid colon staple site in three axes (anterior-posterior, lateral, and cranial-caudal) compared to simulation CT

SECONDARY OUTCOMES:
Intrafraction sigmoid colon organ motion | 90 days
  Offset of the sigmoid colon staple site in three axes (anterior-posterior, lateral, and cranial-caudal) between pre-treatment cone beam computed tomography (CBCT) and post-treatment CBCT
Setup errors | 90 days
  Offset of couch (set-up error) when matching the pre-treatment CBCT with simulation CT

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hung Tsai, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No